CLINICAL TRIAL: NCT03858985
Title: Vagal Nerve Stimulation to Probe Inflammation and Brain in Post-traumatic Stress
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D2920-W
Record Dates: First submitted 2019-02-13; First posted 2019-03-01 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Post-traumatic Stress

STUDY DESIGN:
Intervention Model Description: A sham and active non-invasive vagus nerve stimulator (nVNS) will be used. Both sham and active produce reliable sensation on subject skin over the cervical neck area. The sham device is identical in appearance to the nVNS device. Both devices carry out stimulation for the exact same time period, approximately 2 minutes. Subjects are assigned to sham and nVNS device therapy given once daily for 1 week.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study staff and principle investigator will be blinded to treatment and therefore this study is considered randomized and double blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transcutaneous Vagus Nerve Stimulation (Active Comparator): Cervical Transcutaneous vagus nerve stimulation. Participants will undergo once daily cervical transcutaneous vagus nerve stimulation.
  Interventions: Device: Cervical Transcutaneous Vagus Nerve Stimulation (Active Comparator)
- Sham Vagus Nerve Stimulation (Sham Comparator): Sham Cervical Transcutaneous Vagus Nerve Stimulation. Participants will undergo once daily sham cervical transcutaneous vagus nerve stimulation.
  Interventions: Device: Cervical Transcutaneous Vagus Nerve Stimulation (Sham Comparator)

INTERVENTIONS:
Device: Cervical Transcutaneous Vagus Nerve Stimulation (Active Comparator) — Both sham and active nVNS treatment produce low-voltage electrical signal that induce reliable sensation on subject skin on upper anterior cervical area (overlying carotid artery).
  Arms: Transcutaneous Vagus Nerve Stimulation
Device: Cervical Transcutaneous Vagus Nerve Stimulation (Sham Comparator) — Both sham and active nVNS treatment produce low-voltage electrical signal that induce reliable sensation on subject skin on upper anterior cervical area (overlying carotid artery).
  Arms: Sham Vagus Nerve Stimulation

SUMMARY:
The proposal aims to determine if non-invasive vagus nerve stimulation(nVNS) will alter: 1) the peripheral inflammatory biomarker profile, 2) the neural correlates of change in pain stimuli and 3) PTSD symptom severity and 4) life quality and function in Veterans with PTSD. The planned inflammatory biomarker and neuroimaging results can 1) promote knowledge of inflammatory and neurobiological mechanisms that contribute to pain in PTSD, and 2) advance the ability to provide targeted neuromodulation based interventions that support improved life quality and function for Veterans. These goals are consistent with the VA's mission to sponsor research examining variables related to pathogenesis, diagnosis, and(ultimately) treatment of neuropsychiatric disorders.

DETAILED DESCRIPTION:
Rates of posttraumatic stress disorder (PTSD) are high among combat Veterans with estimates of PTSD within Iraq and Afghanistan Veterans at nearly 17% of active duty and over 24% of reserve service members that screen positive for PTSD. Studies from the current and prior wars have demonstrated that mental disorders, in particular PTSD, are associated with higher rates of: 1) physical symptoms, 2) chronic physical illness and 3) overall mortality. Rates of comorbid PTSD and chronic pain are exceedingly high among Veterans with reports of 30%-50% in both Vietnam and OEF/OIF Veterans, that suggest a shared pathophysiology. Excessive release of peripheral pro-inflammatory cytokines has been implicated in the generation of: 1) pathologic chronic pain states and 2) in PTSD. Perception of an aversive stimulus/threat activates peripheral inflammatory cytokine release, while exogenous administration of an inflammatory stimulus (that also cause release of peripheral inflammatory cytokines) increases the limbic (insular cortex and amygdala) response to aversive/threat stimuli as measured by functional Magnetic Resonance Imaging (fMRI). Work by the investigators' group shows that PTSD influences the: 1) nociceptive response, 2) intrathecal cytokine release and 3) peripheral cytokine release in response to a painful stimulus when compared to responses of Veteran combat controls (CC). Vagus nerve stimulation has been shown to decrease: 1) peripheral inflammatory cytokine release, 2) pain, and 3) anxiety.

Recent work by the group has shown that non-invasive vagal nerve stimulation (nVNS; using extradermal stimulation) decreases peripheral inflammation in healthy control subjects and may similarly decrease hyperinflammation observed in PTSD. In pilot work, the investigators have obtained initial fMRI evidence (preliminary data) suggests that in healthy controls, nVNS decreases insular response to painful stimuli, which is known to be dysregulated in PTSD.

The investigators plan to use nVNS as a probe in PTSD and CC to observe the effects of vagal nerve modulation on: 1) CNS neural circuit function during pain and pain anticipation stimuli, and 2) peripheral inflammatory biomarker measures. The long-term goal of this line of research is to use nVNS as a probe to obtain pilot data of: 1) peripheral inflammatory biomarkers and 2) fMRI derived brain imaging response to pain, to advance the understanding of fundamental pathophysiology of co-morbid pain and PTSD and to ultimately provide, targeted neuromodulation based interventions for Veterans with pain and PTSD. The investigators will study two groups [(PTSD, CC), (both without chronic pain diagnosis)], under two conditions (either nVNS or Sham stimulation), over three time points (pre-nVNS/Sham), (7 days post-nVNS/Sham) and one month after treatment (one month post VNS/Sham). The first objective of this proposal, is to measure peripheral inflammation in response to nVNS treatment in order to delineate peripheral inflammation based biomarker profiles of treatment responsiveness to nVNS in PTSD and CC. The second step is to measure brain region response to a pain and pain anticipation stimuli task before and after nVNS treatment in order to demonstrate: 1) a neural profile of treatment responsiveness to nVNS and 2) the neural profile of nVNS effects on pain in PTSD and CC. Participants will receive a 7-day long nVNS/Sham trial where inflammatory biomarkers, neuroimaging tools, PTSD symptom severity and functional life quality will be assessed before and after the 7 days. Additionally, PTSD symptom severity and functional life quality will be assessed one month after study onset. The direct contrast of pre and post nVNS/Sham will provide an objective and sensitive assessment of neuromodulation with nVNS and lay the groundwork for further neuromodulation based study in PTSD. Such outcomes may provide additional evidence of potential treatment efficacy, thus ultimately provide therapies that enhance VA clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 21 and 65 years, any race or ethnicity.
* For PTSD: Previously deployed, experienced a traumatic event, and meets Clinician-Administered PTSD Scale for DSM-5(CAPS-5) symptom cluster severity criteria for PTSD diagnosis, as well as CAPS total cut-off score > 33. 3. For CC: Previously deployed, experienced a traumatic event, and fails to meet CAPS-5 symptom cluster severity criteria for PTSD diagnosis with CAPS total cut-off score < 20.
* Capable of complying with study schedule, procedures, and speaks English.
* Able to provide voluntary written informed consent prior to initiation of Visit 1; and be able to commit to the return visit at the end of the study.

Exclusion Criteria:

* Rule out significant mental illness, e.g. psychosis, bipolar disorder as well as major depression pre-dating PTSD, based on Structured Clinical Interview for DSM-5(SCID) interview.
* At risk for suicide or homicide(based upon Columbia Suicide Risk Severity Scale(C-SSRS) or BDI-2 screen and follow-up clinical interview).
* Any subject who has undergone evidence-based treatment(CPT or PE) within one month prior to study enrollment or plans to undergo CPT or PE during the study.
* History of head trauma involving loss of consciousness>1 minute and post-concussive symptoms(PCS).
* Chronic pain as defined by pain persisting beyond its ecological alerting function, and clinically defined as lasting longer than 3 months, and/or currently under the care of a chronic pain physician.
* Any condition or therapy that, in the opinion of the investigator and research team, may be significantly worsened by the administration of study treatment or is likely to interfere with the successful collection of the measures required.
* Clinically significant uncontrolled/unstable medical illness or clinically significant surgery within 1 month of the screening visit.
* Evidence of a maladaptive pattern of alcohol use or abuse(based on AUDIT-C interview) one month prior to the screening visit and or illicit drug use or abuse as measured by urine screen positive for illicit substances at the screening Visit 1 or follow up Visit 2.
* Participation in a pharmaceutical trial or exposure to investigational drugs within 1 month of the screening visit.
* Standard of care medications used to treat PTSD will be continued. Any subject that takes anti-inflammatory medications for chronic medical conditions or takes other medications for chronic pain will be excluded.
* MRI-related exclusion criteria: A cardiac pacemaker; metal fragments in eyes/skin/body(shrapnel), subjects who have ever been metal workers/welders; history of eye surgery/eyes washed out because of metal, aortic/aneurysm clips, prosthesis, bypass surgery/coronary artery clips, hearing aid, heart-valve replacement, subjects with an intrauterine device, a shunt(ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators; vision problems uncorrectable with lenses; claustrophobia; inability to lie still on their backs for approximately 60 minutes; prior neurosurgery; or unwillingness or inability to remove nose, ear, tongue, or face rings. Any implants will be reviewed for safety.
* Vagus nerve stimulation related criteria: history of carotid endarterectomy, severe carotid artery disease[e.g. bruits on physical exam or history of transient ischemic attack(TIA) or stroke], congestive heart failure(CHF), cardiac arrhythmia, known severe coronary artery disease or recent myocardial infarction(within 5 years), or a history or seizure or syncope(within the last 1 year), or prior neck surgery will be excluded.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — No women will be enrolled in this study. Prior research suggests that inflammation is sex dependent in individuals with PTSD while inflammation-induced alteration of brain response is also sex specific. There is a known sex difference in the prevalence of PTSD, suggesting that gender may play a role in the pathophysiology of PTSD. Gender differences have repeatedly been shown in human experimental pain paradigms. Taken together only male subjects will be enrolled to decrease variability in measures of pain and peripheral inflammation that could also have sex specific correlation fMRI brain response. If significant effects are demonstrated with this study follow up grant proposals will include female subjects
Enrollment: 88 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Neural Effects Measured by Functional MRI | Functional Imaging Brain Response Measured with Functional MRI: [Time Frame: baseline to week 1 of 1x daily treatment)]
  Examining fMRI derived hemodynamic response curve during rest and pain challenge carried out at baseline to week 1 of 1x daily treatment.
Peripheral Blood Inflammatory Cytokine Measurement | Peripheral Blood Inflammatory Cytokine Measurement: [Time Frame: baseline to week 1 of 1x daily treatment)]
  Peripheral Blood will be drawn to examine concentrations of plasma cytokines in response to sham or nVNS. Cytokine concentrations are measured with in tube whole blood culture system. Peripheral blood cytokine concentration will be quantified in picogram/milliliter.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale | Clinician Administered PTSD Scale: [Time Frame: baseline to week 1 of 1x daily treatment)]
  This semi-structured interview is designed to measure posttraumatic stress disorder diagnostic status as well as symptoms severity. Total scores range from 0 to 20 with higher scores indicating greater severity; change over time will be evaluated.
Sheehan Disability Scale (SDS) | Sheehan Disability Scale (SDS): [Time Frame: baseline to week 1 of 1x daily treatment and post treatment week 5)]
  The Sheehan Disability Scale (SDS) was developed to assess functional impairment in three inter-related domains: work/school, social and family life. It utilizes a 10 point visual analog scale that incorporates spatiovisual, numeric and verbal descriptive anchors to simultaneously assess disability.
WHODAS 2.0 | WHODAS 2.0: [Time Frame: baseline to week 1 of 1x daily treatment and post treatment week 5)]
  The WHODAS 2.0 was developed to assess functional impairment and possesses strong psychometric properties and provides a global disability score as well as six domain scores: cognition, mobility, self-care, getting along with others, participation in society, and life activities. Scores change over time will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Imanuel R Lerman, MD MSc, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No